CLINICAL TRIAL: NCT05140863
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, 12-Week, Phase 3 Study to Evaluate the Efficacy and Safety of HSK16149 Capsules in Chinese Patients With Postherpetic Neuralgia
Brief Title: To Evaluate the Efficacy and Safety of HSK16149 Capsule in Chinese Patients With Postherpetic Neuralgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK16149-302
Record Dates: First submitted 2021-10-14; First posted 2021-12-02 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSK16149 20mg BID (Experimental): HSK16149 20mg, orally twice a day for 12 weeks
  Interventions: Drug: HSK16149 20mg BID
- HSK16149 40mg BID (Experimental): HSK16149 40mg, orally twice a day for 12 weeks
  Interventions: Drug: HSK16149 40mg BID
- Placebo BID (Placebo Comparator): placebo, orally twice a day for 12 weeks
  Interventions: Drug: Placebo BID

INTERVENTIONS:
Drug: HSK16149 20mg BID — HSK16149 20mg, orally twice a day, treatment period; 12-weeks fixed dose
  Arms: HSK16149 20mg BID
Drug: HSK16149 40mg BID — HSK16149 40mg, orally twice a day, treatment period; 12-weeks fixed dose
  Arms: HSK16149 40mg BID
Drug: Placebo BID — Placebo, orally twice a day, treatment period; 12-weeks fixed dose
  Arms: Placebo BID

SUMMARY:
Investigate the Efficacy and Safety of HSK16149 capsules in Chinese Postherpetic Neuralgia Following 12 Weeks Treatment in Comparison to Placebo

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent;
2. Males or females aged 18-75 years of age inclusive;
3. Outpatient, Patients can not stay in the hospital overnight;
4. Patients must have pain present for more than 1 months after the healing of the herpes zoster skin rash;
5. At Screening, pain scale (VAS) of ≥40 mm;

Exclusion Criteria:

1. Peripheral neuropathy or pain unrelated to PHN that may confuse the assessment of PHN;
2. Skin conditions in the area affected by neurupathy that could alter sensation;
3. Chronic systemic diseases that may affect subjects' participation in the study;
4. Severe hematologic, hepatic or renal dysfunction, the subject will be excluded if:1)Neutrophils < 1.5 × 109/L, or platelet < 90 × 109/L, or hemoglobin < 100 g/L, or 2)AST/ALT > 2.5 × upper limit of normal (ULN), or TBIL > 1.5 × ULN, or 3)Estimation of glomerular filtration rate (eGFR) < 60 mL/min / 1.73 m2, or 4)Creatine kinase > 2.0 × ULN.
5. Uncontrolled diabetes(HbA1c≥11.0% at screening) ;
6. History of substance abuse or alcohol abuse;
7. Any active infections at screening;
8. HBsAg or HCV Ab positive, or HIV Ab positive, or serum TP Ab positive;
9. Inability or unwillingness to discontinue any other prohibited concomitant medications (see Section 6.3);
10. Patients who have undergone neurolytic or neurosurgical therapy 1 week before screening for postherpetic neuralgia;
11. Failure to response to previous treatment with pregabalin at doses ≥ 300 mg/d or gabapentin at doses ≥ 1200 mg/d for treatment of PHN;
12. History of allergic or medically significant adverse reaction to investigational products or their excipients, acetaminophen or related compounds;
13. History of suicidal behavior or attempted suicide;
14. Pregnant or preparing for pregnancy or breastfeeding during the study period, or subjects were not willing to use reliable contraceptives methods from the date of ICF signature until 28 days after the last trial drug administration, or planning to use progesterone contraceptives during this period;
15. Mechanical operators who are engaged in high-altitude operations, motor vehicle driving and other dangerous machinery operators;
16. Participated in another clinical study within 30 days prior to screening;
17. Other conditions unlikely to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Compare the change from baseline in ADPS between HSK16149 and placebo at week 12 | Baseline and week 12
  The mean change in average daily pain score (ADPS) was measured using a 11-point numeric rating scale (NRS; 0 [no pain] to 10 [worst possible pain]. The rating averaged over a 7-day period and was based on entries in patients' daily pain diaries

SECONDARY OUTCOMES:
Compare the response rate between HSK16149 and placebo at week 12 (Proportion of subjects whose ADPS decreased by ≥30% and ≥50% from baseline ) | Baseline and week 12
  Ratio of Participants Responding to Treatment, as Measured by Average Daily Pain Score (ADPS) Reduction from Baseline. The ADPS is used to determine categorical response rates.
Compare the change from baseline in ADPS between HSK16149 and placebo at week 1 to 12 | From week 1 to week 12
  The mean change in average daily pain score (ADPS) was measured using a 11-point numeric rating scale (NRS; 0 [no pain] to 10 [worst possible pain]. The rating averaged over a 7-day period and was based on entries in patients' daily pain diaries
Compare the change from baseline in Visual Analogue Scale（VAS） between HSK16149 and placebo at week 12 | Baseline and week 12
  VAS, in which the participant rates pain on a 100 mm-long horizontal line, where 0 mm = no pain and 100 mm = worst possible pain
Compare the change from baseline in Short Form McGill Pain Questionnaire (SF-MPQ) between HSK16149 and placebo at week 12 | Baseline and week 12
  Participants rate their pain in three parts of the questionnaire, which are combined into a single pain intensity score:
  Part 1 - fifteen descriptors of pain intensity, on a scale of 0 (none) to 3 (severe)
  Part 2 - a visual analog scale (VAS), in which the participant rates pain on a 100 mm-long horizontal line, where 0 mm = no pain and 100 mm = worst possible pain
  Part 3 - a Present Pain Intensity index in which the participant rates present pain intensity on a scale of 0 (no pain) to 5 (most intense pain)
Compare the change from baseline in Average Daily Sleep interference score（ADSIS） between HSK16149 and placebo at week 12 | Baseline and week 12
  he sleep interference scores on a scale of 0-10, where 0 = pain did not interfere with sleep to 10 = pain completely interfered with sleep. The weekly ADSIS is based on participants daily sleep interference scores
Compare the total consumption of Acetaminophen and Paracetamol and Dihydrocodeine Tartrate between HSK16149 and placebo during the trial | From week 1 to week 12
Compare the change from baseline in EQ-5D-5L between HSK16149 and placebo at week 12 | Baseline and week 12
  The change from baseline in total EuroQol-5-Domain-5-Level health questionnaire
AE（adverse event） to evaluate the safety of HSK16149 during the trial | From week 1 to week 12
  Number and severity of AEs
Peak Plasma Concentration (Cmax) of HSK16149 capsules in Chinese patients with Postherpetic Neuralgia | Week 4,week 8,week 10,week 12
Area under the plasma concentration versus time curve (AUC) of HSK16149 capsules in Chinese patients with Postherpetic Neuralgia | Week 4,week 8,week 10,week 12

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Dermatology Hospital of Chinese Academy of Medical Sciences, Nanjing, Jiangsu
  - The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi

REFERENCES:
- [Derived] Zhang D, Lei T, Qin L, Li C, Lin X, Wang H, Zhang G, Zhang S, Shi K, Li L, Yang Z, Yang X, Ba X, Gao Y, Zhang Z, Wang G, Wu L, Wang Y, Wang Y, Zhu S, Shi J, Ye Z, Yang C, Liu C, Zhang T, Lu S, Yu N, Li X, Han X, Chen X, Wan L, Cheng Z, Bai N, Jin Z, Yu C, Zhang W, Lu J, Wang D, Sun H, Wu W, Qin P, Feng Z, Chen R, Zhang T, Yang D, Yin W, Zhang J, Li X, Li F, Wu T, Lu Q. Efficacy and Safety of Crisugabalin (HSK16149) in Adults with Postherpetic Neuralgia: A Phase 3 Randomized Clinical Trial. JAMA Dermatol. 2024 Nov 1;160(11):1182-1191. doi: 10.1001/jamadermatol.2024.3410. PMID 39320907